CLINICAL TRIAL: NCT05859347
Title: Development of a Novel, Scalable, Neurobiologically-Guided Transcranial Magnetic Stimulation Protocol for the Treatment of Cannabis Use Disorder
Brief Title: Repetitive Transcranial Magnetic Stimulation for Cannabis Use Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Brain & Behavior Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-233
Record Dates: First submitted 2023-04-11; First posted 2023-05-16 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Cannabis Use Disorder
Keywords: Repetitive Transcranial Magnetic Stimulation; Cannabis; Substance Use Disorder; Prefrontal Cortex; Insula; Neuroimaging
MeSH Terms: conditions — Marijuana Abuse; Substance-Related Disorders | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of two groups to receive either high-frequency (10 Hz) or low-frequency (1 Hz) rTMS.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-Frequency (HF) (Active Comparator): 10 Hz rTMS
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation
- Low-Frequency (LF) (Active Comparator): 1 Hz rTMS
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation — rTMS is a non-invasive neuromodulatory technique that applies alternating magnetic fields to the scalp to induce electric currents in localized cortical tissue. The intervention (LF or HF rTMS) will be administered daily 5 days/week for 4 weeks, using the MagVenture MMC-140 circular coil, with the brain regions targeted as the bilateral prefrontal cortex and the insula.
  Other Names: MagVenture MMC-140 Coil

SUMMARY:
There has been a considerable rise in cannabis consumption in recent years, with estimates of 200 million individual users globally. Importantly, 3% of these individuals have cannabis use disorder (CUD), with this prevalence increasing to 33% amongst regular users, making it one of the most common substances use disorders (SUDs) worldwide. CUD is associated with substantial health, societal, and economic costs, and worsening of other psychiatric disorders. Despite this clinical burden, effective treatment options are limited. No pharmacological treatments have emerged as clearly efficacious, and psychotherapeutic interventions have shown tempered results.

Repetitive transcranial magnetic stimulation (rTMS) is a non-invasive brain-based approach in which alternating magnetic fields are applied to the scalp to induce electrical currents in cortical tissue. As it can modulate neural circuits implicated in neuropsychiatric disorders, it is a promising brain-based approach in the treatment of addictions. Evidence has indicated its efficacy in reducing drug craving and consumption across numerous SUDs, although research into cannabis has been largely unexplored. Recently, a novel circular rTMS coil, the MagVenture MMC-140, has been developed with the capacity to modulate both the bilateral prefrontal cortex (PFC) and insula, both of which are implicated in the neurocircuitry of craving and executive function. As such, it shows potential for CUD treatment.

This proof-of-concept clinical trial will evaluate the feasibility and tolerability of a 4-week course of rTMS to the PFC/insula using MMC-140 as a treatment for CUD. Feasibility of both high frequency (HF; excitatory) and low frequency (LF; inhibitory) stimulation parameters will be evaluated. In addition, pre/post rTMS changes in cannabis use outcomes (e.g., consumption, craving, and withdrawal), executive function, and PFC/insula functional connectivity will be explored. By comprehensively investigating clinical, cognitive, and neuroimaging effects of rTMS, this study could pave the way for the first brain-based intervention in CUD that could be widely adopted into clinical settings using a novel, cost-effective and accessible rTMS device.

ELIGIBILITY:
Inclusion Criteria:

1. Must be deemed to have capacity to provide informed consent
2. Age between 18 to 65
3. Diagnosis of cannabis use disorder according to the DSM-5 and the Structured Clinical Interview for DSM-5 (SCID for DSM-541)
4. Report cannabis as the primary drug of concern, a frequent pattern of use (≥5 days per week), and a goal of reduction or abstinence of cannabis use
5. CUDIT-R score ≥12
6. Marijuana Contemplation Ladder ≥7
7. Cannabis positive urine drug screen, with Narcochek baseline THC-COOH level of >150 ng/ml.
8. On a stable regimen of their psychotropic medications for 14 days before enrolment.

Exclusion Criteria:

1. Pregnant or intending to be pregnant during the study
2. Diagnosis of bipolar disorder, schizophrenia spectrum disorder, or other active concurrent psychiatric disorder that is too unstable and may preclude safe participation in the trial as deemed by the PI.
3. Substance use disorder other than cannabis or nicotine, that is of moderate severity or greater, or is the primary substance of concern based on the SCID for DSM-5
4. Known active seizure disorder, significant head injury with an imaging verified lesion
5. Unstable medical illness
6. Presence of cardiac pacemaker, intracranial implant, or metal in the cranium
7. Participants taking > 2 mg lorazepam (or a benzodiazepine at an equivalent dose) or taking any anticonvulsant medication during treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Feasibility of study completion as assessed by completion rates | The timeframe is through study completion, beginning from baseline to end of rTMS treatment week 4, an average of 8 weeks, the event determined by withdrawal from the study.
  Feasibility is determined by completion of the study and all associated study assessments, without withdrawing or being withdrawn from the study. Withdrawal from the study can be dropping out for any reason, including intolerability, serious adverse events, or inability to adhere to study procedures.
Tolerability of Intervention as assessed by adverse event reporting | The timeframe is through study completion, beginning from baseline to end of rTMS treatment week 4, an average of 8 weeks. The events being counts of adverse events or serious adverse events.
  This will be assessed through a side effect report at each treatment session. Safety monitoring will be implemented through the documentation and monitoring of adverse events (AEs) and serious adverse events (SAEs) using incidence tables by severity, relationship to treatment and baseline parameters.

SECONDARY OUTCOMES:
Cannabis Use | Baseline (pre-rTMS), Weekly (end of each week of rTMS), Follow-up (4-weeks post-rTMS), up to a total time frame of 8 weeks. Events are counted as self reported instances of cannabis use on the Timeline Followback.
  Determined through self-report on the Timeline Followback (TLFB). Endpoints of interest will include percentage of days per week using cannabis, number of use sessions per day, 7-day point prevalence abstinence. Semi-quantitative analysis of cannabis use will be obtained through a THC Pre-Dosage Test (Narcocheck ®, Villejuif, France) to confirm.
Cannabis Craving | Baseline (pre-rTMS), Weekly (end of each week of rTMS), an average of 8 weeks from baseline assessment to end of rTMS, Follow-up (4-weeks post-rTMS),
  Changes in cannabis craving assessed through the Marijuana Craving Questionnaire (MCQ). Minimum score is 3 and maximum score is 84. Higher scores indicate greater cannabis craving (worse outcome).
Cannabis Withdrawal | Baseline (pre-rTMS), Weekly (end of each week of rTMS), an average of 8 weeks from baseline assessment to end of rTMS, Follow-up (4-weeks post-rTMS),
  Changes in cannabis withdrawal symptoms assessed through the Marijuana Withdrawal Checklist (MWC)
Prefrontal cortex and Insula Connectivity | Baseline (pre-rTMS), End of rTMS (end of treatment week 4 of rTMS)
  Assessed by seed-based resting state connectivity on functional magnetic resonance imaging (fMRI). Seeds are defined as the medial prefrontal cortex, dorsolateral prefrontal cortex, and the insula. Measurement will be of change in strength of connectivity between these seeds pre- to post-rTMS, and comparing between groups (high or low frequency stimulation).
Depression symptoms | Baseline (pre-rTMS), Weekly (end of each week of rTMS), an average of 8 weeks from baseline assessment to end of rTMS, follow-up (4-weeks post-rTMS),
  Changes in depression symptoms assessed through the 17-item Hamilton Rating Scale for Depression (HRSD-17). Minimum score is 0, maximum score is 52, higher scores indicate greater depression (worse outcome)
Anxiety symptoms | Baseline (pre-rTMS), Weekly (end of each week of rTMS), an average of 8 weeks from baseline assessment to end of rTMS, follow-up (4-weeks post-rTMS),
  Changes in anxiety symptoms assessed through the Generalized Anxiety Disorder Scale 7 (GAD-7). Minimum score is 0, maximum score is 21, higher scores indicate greater anxiety (worse outcome).
Trail Making Test | Baseline (pre-rTMS), End of rTMS (end of treatment week 4 of rTMS), an average of 8 weeks from baseline assessment to end of rTMS, follow-up (4-weeks post-rTMS)
  Changes on a neuropsychological assessment for attention, speed, and mental flexibility. Part A and Part B. Measurement: number of seconds required to complete the task. • Higher scores reveal greater impairment.
Digit Span | Baseline (pre-rTMS), End of rTMS (end of treatment week 4 of rTMS), an average of 8 weeks from baseline assessment to end of rTMS, follow-up (4-weeks post-rTMS)
  Changes on a neuropsychological assessment for working memory. Consists of 2 parts: Forwards and Backwards. Each item is scored 0, 1, or 2 points. (Depending on accuracy). • Lower scores reveal greater impairment. Minimum score 0. Maximum total score on Digit Span: 30 points
Hopkins Verbal Learning Test | Baseline (pre-rTMS), End of rTMS (end of treatment week 4 of rTMS), an average of 8 weeks from baseline assessment to end of rTMS, follow-up (4-weeks post-rTMS)
  Changes on a neuropsychological assessment for working memory. Consists of 3 parts: A (free recall), B (delayed recall), C (recognition). Less number of words remembered indicates worse outcome.
Continuous Performance Test | Baseline (pre-rTMS), End of rTMS (end of treatment week 4 of rTMS), an average of 8 weeks from baseline assessment to end of rTMS, follow-up (4-weeks post-rTMS)
  Changes on a neuropsychological assessment for sustained attention. Measurement & Scoring Categories: Correct Detection (number of times the client responded to the target stimulus. Higher rates of correct detections indicate better attentional capacity), reaction times (Amount of time between the presentation of the stimulus and the client's response), omission errors (Number of times the target was presented, but the client did not respond/click the mouse. High omission rates indicate distractibility to stimuli or a sluggish response), commission errors (Number of times the client responded but no target was presented. A fast reaction time and high commission error rate points to difficulties with impulsivity. A slow reaction time with high commission and omission errors, indicates inattention in general).

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada